CLINICAL TRIAL: NCT00686569
Title: Mediastinal Microdialysis in Early Diagnosis of Anastomotic Leakage After Resection for Esophageal Cancer: Preliminary Results
Brief Title: Mediastinal Microdialysis in Patients With Oesophageal or Cardia Cancer Treated by Resection
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Niels Qvist, Professor, Odense University Hospital
Other Study IDs: S-20070062
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Anastomotic Leakage; Esophageal Cancer
MeSH Terms: conditions — Anastomotic Leak; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Postoperative anastomotic leakage is a serious complication in patients with oesophageal or cardia cancer. Early diagnosis and treatment are mandatory. The primary aim of the present study is to investigate the clinical use of mediastinal microdialysis and whether is able to detect anastomotic leakage prior to the development of clinical symptoms.

DETAILED DESCRIPTION:
Patients undergoing oesophageal or cardia resection for cancer are monitored by mediastinal microdialysis during the postoperative period. Subcutaneous microdialysis serves as a control. Samples are collected every 4-hour. Samples will be analyzed continuously but the results will not be included in the clinical evaluation of the patient.

A total of 30 patients will be included in this pilot study. The results of the mediastinal microdialyses will be compared with the clinical course in each patient. The results form the uncomplicated courses will be used to define the normal variations in mediastinal microdialysis. This will be compared to results from patients with various complications.

ELIGIBILITY:
Inclusion Criteria:

* Histological verified oesophageal or cardia cancer

Exclusion Criteria:

* Lack of consent, otherwise none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoin oesophageal resection for cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Early detection of postoperative complications | 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Niels Qvist, Professor, Study Chair — Department of Surgery
Locations (2):
- Denmark (2):
  - Surgical department A, Odense University Hospital, Odense
  - Odense University Hospital, surgical department A, Odense C

REFERENCES:
- [Result] Ellebaek M, Qvist N, Fristrup C, Mortensen MB. Mediastinal microdialysis in the diagnosis of early anastomotic leakage after resection for cancer of the esophagus and gastroesophageal junction. Am J Surg. 2014 Sep;208(3):397-405. doi: 10.1016/j.amjsurg.2013.09.026. Epub 2014 Jan 16. PMID 24656920